CLINICAL TRIAL: NCT00150683
Title: Evaluation of Conventional and Innovative Standing Frame for the Treatment of Osteoporosis After Spinal Cord Injury
Brief Title: Effectiveness of Vibration and Standing Versus Standing Alone for the Treatment of Osteoporosis for People With Spinal Cord Injury.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Ontario Neurotrauma Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONBO-99135; Ontario Neurotrauma Foundation
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2005-09-08 (Estimated); Status verified 2005-09

CONDITIONS: Spinal Cord Injury.; Osteoporosis.
Keywords: Spinal Cord Injury.; Osteoporosis.; Standing.; Vibration.
MeSH Terms: conditions — Spinal Cord Injuries; Osteoporosis

INTERVENTIONS:
Device: vibration and passive standing versus passive standing alone

SUMMARY:
The purpose of this study is to find out if standing and/or standing with vibration works for the treatment of osteoporosis for people with a spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic spinal cord injury of greater than 12 months.
* Osteopenia or osteoporosis of the hip.

Exclusion Criteria:

* Pregnant or lactating females.
* Nonunion lower extremity fracture within the last 6 months.
* Bilateral hip or knee flexion contractures.
* Bilateral lower extremity total hip or knee replacement.
* Heterotopic ossification of the hip or knee.
* Concurrent treatment with a bisphosphonate.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1999-03; Study Completion 2001-07

PRIMARY OUTCOMES:
Change in bone mineral density from baseline of the hip, distal femur and proximal tibia at 6-months and 12-months.

SECONDARY OUTCOMES:
Spasticity (modified Ashworth).
Quality of life.
Frequency and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: B. Cathy Craven, BPHE, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehab, Lyndhurst Centre, Toronto, Ontario, Canada